CLINICAL TRIAL: NCT04749693
Title: Observational Study of the Use of DBLG1 System in Real Life
Acronym: SP12
Status: Recruiting | Type: Observational
Sponsor: Diabeloop (Industry)
Responsible Party: Sponsor
Other Study IDs: RCB 2020-A 02808-31
Record Dates: First submitted 2021-02-02; First posted 2021-02-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Type1diabetes
Keywords: Type 1 Diabetes; HbA1c > 8%; Closed loop system; insulin pump; Algorithm; Real life
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with HbA1c >= 8% despite the use of insulin pump and frequent glycemic control: only group included in the study
  Interventions: Device: DBLG1 System

INTERVENTIONS:
Device: DBLG1 System — Use of DBLG1 System in real life condition

SUMMARY:
This study will be conducted on human subjects and is observational, prospective and uncontrolled, defined as a category 3 according to the Jardé Law (RIPH3). It is a national and multicentric study. Enrolled patients are Type 1 Diabetes (T1D) patients who receive the DBLG1 System (CE marked medical device) to be treated. Patients have their regular visits with their own clinician. No change from their usual care must and will be done, including trainings and treatment. At the end of the study, patients will keep their system for their usual care and will continue having usual follow-up visits with their clinician.

Data related to their glycemia, complications and quality of life will be collected for 1 year from the beginning of their treatment. A comparison with data collected during the 2 weeks of run-in period, prior to the activation of loop mode, is planned. In case the run-in phase lasts longer than 2 weeks, data collected from the two last weeks only will be kept for analysis and comparison.

The study is completed when all patients have their "end of study" file completed in the electronic Case Report Form (eCRF).

DETAILED DESCRIPTION:
The study is designed to address the specific requirements from National Commission for the Evaluation of Medical Devices and Health Technologies (CNEDiMTS) and to complete data obtained up to now, with a larger cohort and in real life settings.

In order to increase variability in the profiles of patients included and to be as representative as possible of all eligible patients, 20 centers will participate in the study, both private and public, with a mix of university and regional centers and 348 patients will be included consecutively.

The inclusion period lasts 6 months and each patient will be included in the study for a period of 2 weeks of run-in and 1 year of treatment. An inclusion period of 6 months is enough according to investigation site data and estimation of inclusion over 6 months (detailed in part Healthcare professional and investigation centers recruitment).

This study is observational. Patients included follow their usual medical care and will only be asked for the specific need of the study to answer two questionnaires (at the beginning and at the end of the study) and give their HbA1c results performed in their current medical follow-up. As it is a post-registration study, medical devices are provided to patients on medical prescription by healthcare providers, which have signed a distribution agreement with and have been trained by Diabeloop. Patients have their system for 4 a maximum of 4 years (life duration of the medical device (DBLG1 System)).

Patients follow-up visits are not mandatory and no frequency is imposed. Investigators, according to their habits, have follow-up visits corresponding to what they usually propose to patients having a new treatment.

During the whole study and apart from scheduled visits (inclusion, beginning of run-in, beginning of treatment , enf of study), each patient may contact his/her clinician investigator in case of issue he/she judges as serious, for questions, etc. In that case, the clinician may program a visit with the patient and deal with adverse events. Phone calls are recorded in Case Report Form (CRF), as well as on-site visits.

Note: with Yourloops; investigators may follow the state of their patients, regarding the time in range, mean glycemia value etc. Based on this, they may require a visit at their convenience with the patient in order to change parameters of the system, discuss adverse events, etc.

Objectives are the following To evaluate improvement in blood glucose control with use of DBLG1 System after one year in real life.

To evaluate details of glycemic control improvement, safety and adverse events due to the DBLG1 System, evolution of quality of life after one year in real life and healthcare professional support.

Study endpoints Improvement of the time in glycemic range 70 - 180 mg/dL, in percentage, on 24hours and nighttime.

HbA1c Mean CGM glucose - on 24hours and nighttime Time in 70 - 140 mg/dL range on 24hours and nighttime only Time in hypoglycemia (under 70 mg/dL, 60 mg/dL and 50 mg/dL) - on 24hours and nighttime Time in hyperglycemia (above 180 mg/dL, 250 mg/dL and 300 mg/dL) - on 24hours and nighttime Percentage of time using activated loop mode vs. deactivated loop mode Standard Deviation (SD) and Coefficient of variation (CV) of Continuous Glucose Monitoring (CGM) values on 24hours and nighttime Number and type of adverse events Overall and diabetic-specific quality of life Quantification of the healthcare professional support required

An descriptive interim analysis will be made on the first 100 enrolled patients after 6 months of use of the DBLG1.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 diabetes;
* patients who are at least 18 years old;
* patients total daily dose required must be less than 90 units (U);
* patients accepting to be treated with 100 U/mL rapid-acting insulin analog
* patients having a HbA1c ≥ 8% despite of the use of a pump for at least 6 months
* patients performing glucose self-monitoring several times ( ≥ 4) a day
* patient accepting the technology
* patients agreeing to use the system with activated loop mode during at least 75% of the
* total time of use, this will be analyzed after 1 year of use.
* patients must be affiliated to any kind of social security

Exclusion Criteria:

* patients receiving a total daily dose of insulin lower than 8 U;
* patients suffering from a serious illness or having a treatment that might significantly impair diabetes physiology (iSGLT2, steroids, metformin), i.e. glucose-insulin interactions, that might interfere with the medical device (for example treatment by steroids with variable dosage during the study period);
* patients having severe uncorrected problems of hearing and/or visual acuity preventing proper use of DBLG1 System;
* patients unable to understand and perform all of the instructions regarding the devices and the clinical investigation provided by Diabeloop.
* patients planning to perform during the year of study repeated magnetic resonance imaging (MRI), computed tomography (CT) scan, or high-frequency electrical heat (diathermy) treatment. The G6 has not been tested in those situations. The magnetic fields and heat could damage the components of the Dexcom G6, which may cause it to display inaccurate sensor glucose readings (readings) or may prevent alerts. Without G6 readings or alarm/alert notifications, patients might be exposed to severe low or high glucose events;
* patients who are unwilling or unable to maintain contact with the healthcare professional;
* patients willing to use any insulin that is not 100 U/mL rapid-acting insulin analog with the system (for example regular insulin; long-acting insulin analog; 200 U/mL rapid-acting insulin analog)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type 1 diabetes equal or more than 18 years old, with Hb1Ac ≥ 8%
Sampling Method: Non-Probability Sample
Enrollment: 348 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
time in 70 - 180 mg/dL glycemic range | through study completion, an average of 1 year
  Improvement of the time in glycemic range 70 - 180 mg/dL, in percentage, on 24hours and nighttime

SECONDARY OUTCOMES:
HbA1c HbA1c HbA1c | at the beginning and at the end of the study (1 year between each value)
  change in the HbA1c after 1 year of use of the device
mean CGM | through study completion, an average of 1 year
  change of mean CGM glucose on 24hours and nighttime
time in 70 - 140 mg/dL glycemic range | through study completion, an average of 1 year
  change of time in 70 - 140 mg/dL range on 24hours and nighttime
time in hypoglycemia | through study completion, an average of 1 year
  change of time in hypoglycemia, under 70 mg/dL, 60 mg/dL and 50 mg/dL on 24hours and nighttime
time in hyperglycemia | through study completion, an average of 1 year
  change of time in hyperglycemia above 180 mg/dL, 250 mg/dL and 300 mg/dL on 24hours and nighttime
use of loop mode | treatment period, an average of 1 year
  percentage of time using activated loop mode vs. deactivated loop mode
SD and CV of CGM values | through study completion, an average of 1 year
  change of SD and CV of CGM values on 24hours and nighttime
adverse event | through study completion, an average of 1 year
  number of adverse events
Health Survey | at the beginning and at the end of the study (1 year between each value)
  change of the patient health, evaluated by questionnaire Short Form 12 Health Survey filled in at the beginning and at the end of the study
Fear of hypoglycemia | at the beginning and at the end of the study (1 year between each value)
  change of the patient fear of hypoglycemia, evaluated by questionnaire Hypoglycemia fear survey filled in at the beginning and at the end of the study
Patient stress status | at the beginning and at the end of the study (1 year between each value)
  change of the patient stress status, evaluated by questionnaire Diabetes distress scale, filled in at the beginning and at the end of the study
Acceptability of the device | at the beginning and at the end of the study (1 year between each value)
  change of the patient's satisfaction of previous vs. DBLG1 System devices, evaluated by questionnaire patient stress status, filled in at the beginning and at the end of the study
incidence of the system on the necessary healthcare professional charge | through study completion, an average of 1 year
  questionnaire at each visit (duration and type of visit, number and type of healthcare professional required for the visit)

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Schaepelynck, Principal Investigator — APHM Hôpital Sud Sainte Marguerite; Lucy Chaillous, Principal Investigator — Nantes University Hospital; Hélène Hanaire, Principal Investigator — University Hospital, Toulouse; Sandrine Lablanche, Principal Investigator — University Hospital, Grenoble; Alfred Penfornis, Principal Investigator — CH Sud Francilien; Yves Reznik, Principal Investigator — CHU CAEN
Locations (20):
- France (20):
  - Hôpital Avicenne APHP, Bobigny
  - Hôpital de la cavale blanche, Brest
  - CHU Caen, Caen
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Bocage Central, Dijon
  - Hôpital Simone Veil, Eaubonne
  - CHU Grenoble, Grenoble
  - Groupe Hospitalier La Rochelle - Ré - Aunis, La Rochelle
  - CHU Lille, Lille
  - Diab-e-Care, Lyon
  - Hôpital Européen, Marseille
  - Hôpital la conception, pole ENDO, Marseille
  - hôpital Nord Laennec, Nantes
  - Lariboisière - Fernand Widal APHP, Paris
  - Hôpital Bichet Claude Bernard - APHP, Paris
  - Clinique Princess, Pau
  - CHU Reims, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpital civil de Strasbourg, Strasbourg
  - Hôpital de Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No